CLINICAL TRIAL: NCT04672486
Title: PRIDE - Pilot Trial of an Online Digital Problem-solving Intervention for School-going Adolescents in Goa, India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sangath (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); University of Sussex (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PG_2020_69; 106919/Z/15/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Mental Health Issue; Depression, Anxiety; Stress
Keywords: digital mental health intervention; adolescent mental health
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A two-arm, individually randomized controlled trial with equal allocation of participants between arms.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants will be offered an online problem-solving intervention that is delivered through a smartphone app (called POD Adventures) with telephone-based guidance from a lay counsellor. The app teaches problem-solving skills through interactive animated vignettes and personalized action plans, with encouraging prompts and feedback offered through an in-app guide character. In addition, methods of gamification are used to model and practice complementary coping strategies (e.g., relaxation) and enhance engagement. Participants will use the app remotely (i.e., from their home) in their own time.
  Interventions: Behavioral: POD Adventures
- Usual Care (No Intervention): Participants randomized to the control arm will be provided with usual care. This will consist of information and contact details about local mental health service providers and two recently established government provided/affiliated helplines: (i) Manodarpan, a student mental health helpline supported by the Ministry of Human Resource Development; and (ii) a 24/7 mental health helpline (KIRAN) supported by the Social Justice and Empowerment Ministry. The same information will be provided to participants in the intervention arm.

INTERVENTIONS:
Behavioral: POD Adventures — Participants in the intervention arm will receive information about local services/national helplines and a brief problem-solving intervention that is delivered through a smartphone app with telephone guidance from a lay counsellor. The intervention is grounded in stress-coping theory, with a technical focus on practical problem solving. The emphasis on problem solving reflects the primacy of psychosocial stressors in adolescent help-seeking. Moreover, problem-solving is among the most commonly used practice elements in evidence-based psychological interventions for children and adolescents globally.
  The content of the app comprises two sections: 'Adventures' which teaches problem-solving concepts and methods through contextually-appropriate games; and 'My POD' which scaffolds the student through the application of step-by-step problem-solving procedures to their own prioritized problems.
  Arms: Intervention Arm

SUMMARY:
This study is part of a Wellcome Trust-funded research programme in India called PRIDE (PRemIum for aDolEscents, 2016-2022) led by Principal Investigator Prof. Vikram Patel (Harvard Medical School). The programme aims to develop and evaluate a trans-diagnostic, stepped-care intervention targeting common mental health problems in school-going adolescents in India.

The study is planned in the context of school closures and other COVID-19 mitigation strategies in India. We will undertake a pilot randomized controlled trial with the specific aims to

* assess the acceptability and feasibility of an online problem-solving intervention
* obtain effect size estimates for the online problem-solving intervention when compared to a usual care control condition
* assess process variables related to intervention and research procedures and thereby assist with planning for a future large-scale trial.

DETAILED DESCRIPTION:
BACKGROUND:

PRIDE has been implemented in India to address the scarcity of evidence-based interventions for common adolescent mental health problems nationally and in low-resource settings more widely. The goal is to develop and evaluate a suite of scalable, transdiagnostic psychological interventions (i.e., suitable for a variety of mental health presentations) that can be delivered by non-specialist ('lay') counsellors in resource-poor school settings. It builds upon India's national initiative for adolescent health, launched in 2014, which emphasises mental health as a public health priority and schools as an important platform for youth-focused treatment delivery.

The development of the PRIDE school-based intervention model has been founded on the principle of stepped care which reserves increasingly specialised, resource-intensive interventions for individuals who do not respond to simpler first-line treatments. Previous PRIDE studies (Parikh 2019, Michelson 2019, Michelson 2020) revealed a high demand for school-based psychological support among socially disadvantaged adolescents. A majority of these adolescents do not meet conventional clinical thresholds for mental disorder, but may still benefit from early intervention to mitigate risks for developing more severe and socially disabling mental health problems in the longer-term.

Hence, the aim of the current study is to evaluate the effectiveness of an online 'open-access' digital intervention for adolescents who have a felt need for psychological support irrespective of assessed psychopathology. Online delivery is necessary due to prevailing COVID-19 restrictions that include school closures and a shift to online schooling for the remainder of the academic year.

SIGNIFICANCE:

This study comprises one of the first online adolescent mental health trials in the context of the COVID-19 outbreak in India. The study will take an existing digital mental health intervention developed and evaluated by our group in India and repurpose this platform for online delivery.

Problem solving was selected as the core intervention component based on global evidence for its generalised (i.e., transdiagnostic) benefits across diverse mental health presentations and its specific relevance to common stressors observed in the target population.

The findings are likely to be generalisable to routine settings since the research will be implemented in government-aided secondary schools which cater to low-income communities. External validity will be further strengthened through idiographic outcome assessment alongside standardised assessment instruments, and broad eligibility criteria which do not exclude any specific mental health presentations.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled as a student in grades 9-12 (ages 13-19 years) at one of the collaborating schools;
* Able to access an Android smartphone with internet and a valid phone number for the six-week duration of the study;
* Wanting psychological help for managing stressful situations or internal states;
* Proficient in written and spoken English, as needed to participate fully in study procedures;
* For adolescents under 18 years of age, provides informed assent to participate, supported by parental consent;
* For adolescents 18 years of age or over, provides informed consent to participate.

Exclusion Criteria:

* Unable to understand intervention materials (for example, due to a reading or hearing disability or inability to comprehend Hindi, Konkani, or English).

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 11 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Youth Top Problems (YTP) | 6 weeks
  The Youth Top Problems (YTP) is a youth-reported idiographic measure of psychosocial problems that identifies, prioritizes and scores adolescents' three main concerns. Each of the nominated concerns is scored from 0 (not a problem) to 10 (huge problem). A mean severity score can be calculated across the nominated problems. It has been translated and used in previous PRIDE studies in consultation with one of the original developers of the measure (Prof. Bruce Chorpita, UCLA).

SECONDARY OUTCOMES:
Revised Child Anxiety and Depression Scale - Short Version (RCADS-25) | 6 weeks
  This is a 25-item questionnaire that assesses for DSM-IV (APA, 2000) related anxiety and depression dimensions in children and adolescents. The measure asks youth to rate how often they experience each item (e.g. "worries that something bad will happen to me") on a 4-point Likert scale ranging from 0 (never) to 3 (always). The RCADS produces a Total Anxiety Scale, which is a sum of five subscales: Generalized Anxiety Disorder, Separation Anxiety Disorder, Social Phobia, Panic Disorder, and Obsessive-Compulsive Disorder. A sixth subscale, Major Depressive Disorder, asks about depressive symptoms. The measure has been used with adolescents in a large number of international studies, including in India (Piqueras 2017, Haldar 2016).

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Patel, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM); Daniel Michelson, PhD, Study Director — University of Sussex
Locations (1):
- Sangath, Goa, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
See below.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after completion of the study
Access Criteria: Access to data will be granted to researchers after review of requests by the PI and in accordance with the guidelines of sponsors, collaborators and the study funder.

REFERENCES:
- [Background] Michelson D, Malik K, Krishna M, Sharma R, Mathur S, Bhat B, Parikh R, Roy K, Joshi A, Sahu R, Chilhate B, Boustani M, Cuijpers P, Chorpita B, Fairburn CG, Patel V. Development of a transdiagnostic, low-intensity, psychological intervention for common adolescent mental health problems in Indian secondary schools. Behav Res Ther. 2020 Jul;130:103439. doi: 10.1016/j.brat.2019.103439. Epub 2019 Jul 30. PMID 31466693
- [Background] Gonsalves PP, Hodgson ES, Kumar A, Aurora T, Chandak Y, Sharma R, Michelson D, Patel V. Design and Development of the "POD Adventures" Smartphone Game: A Blended Problem-Solving Intervention for Adolescent Mental Health in India. Front Public Health. 2019 Aug 23;7:238. doi: 10.3389/fpubh.2019.00238. eCollection 2019. PMID 31508404
- [Background] Gonsalves PP, Hodgson ES, Bhat B, Sharma R, Jambhale A, Michelson D, Patel V. App-based guided problem-solving intervention for adolescent mental health: a pilot cohort study in Indian schools. Evid Based Ment Health. 2021 Feb;24(1):11-18. doi: 10.1136/ebmental-2020-300194. Epub 2020 Nov 18. PMID 33208507
- [Background] Michelson D, Malik K, Parikh R, Weiss HA, Doyle AM, Bhat B, Sahu R, Chilhate B, Mathur S, Krishna M, Sharma R, Sudhir P, King M, Cuijpers P, Chorpita B, Fairburn CG, Patel V. Effectiveness of a brief lay counsellor-delivered, problem-solving intervention for adolescent mental health problems in urban, low-income schools in India: a randomised controlled trial. Lancet Child Adolesc Health. 2020 Aug;4(8):571-582. doi: 10.1016/S2352-4642(20)30173-5. Epub 2020 Jun 23. PMID 32585185
- [Background] Piqueras JA, Martin-Vivar M, Sandin B, San Luis C, Pineda D. The Revised Child Anxiety and Depression Scale: A systematic review and reliability generalization meta-analysis. J Affect Disord. 2017 Aug 15;218:153-169. doi: 10.1016/j.jad.2017.04.022. Epub 2017 Apr 20. PMID 28475961
- [Background] Haldar, Kasturi. (2016). Adapting a Revised Child Anxiety and Depression Scale for rural India: a pilot, amenable to scale up. DoI: 10.31234/osf.io/25pnr.
- [Derived] Gonsalves PP, Sharma R, Hodgson E, Bhat B, Jambhale A, Weiss HA, Fairburn CG, Cavanagh K, Cuijpers P, Michelson D, Patel V. A Guided Internet-Based Problem-Solving Intervention Delivered Through Smartphones for Secondary School Pupils During the COVID-19 Pandemic in India: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2021 Oct 6;10(10):e30339. doi: 10.2196/30339. PMID 34586075